CLINICAL TRIAL: NCT02924818
Title: Cohort for Research and Innovation in Chronic Inflammatory Respiratory Diseases: The RINNOPARI Project
Brief Title: Cohort for Research and Innovation in Chronic Inflammatory Respiratory Diseases
Acronym: RINNOPARI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PO16020*
Record Dates: First submitted 2016-10-04; First posted 2016-10-05 (Estimated); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Chronic Inflammatory Pulmonary Diseases
MeSH Terms: interventions — Surveys and Questionnaires; Respiratory Physiological Phenomena; Hematologic Tests; Shadowing Technique, Histology; X-Rays

ARMS (5):
- Chronic Obstructive Pulmonary disease (COPD) (Experimental)
  Interventions: Other: Clinical assessment; Behavioral: questionnaires; Other: pulmonary function test; Biological: blood test; Biological: microbiology; Biological: histology; Other: imaging
- Cystic Fibrosis (CF) (Experimental)
  Interventions: Other: Clinical assessment; Behavioral: questionnaires; Other: pulmonary function test; Biological: blood test; Biological: microbiology; Biological: histology; Other: imaging
- bronchiectasis (Experimental)
  Interventions: Other: Clinical assessment; Behavioral: questionnaires; Other: pulmonary function test; Biological: blood test; Biological: microbiology; Biological: histology; Other: imaging
- Interstitial lung disease (ILD) (Experimental)
  Interventions: Other: Clinical assessment; Behavioral: questionnaires; Other: pulmonary function test; Biological: blood test; Biological: microbiology; Biological: histology; Other: imaging
- controls (Experimental)
  Interventions: Other: Clinical assessment; Behavioral: questionnaires; Other: pulmonary function test; Biological: blood test; Biological: microbiology; Biological: histology; Other: imaging

INTERVENTIONS:
Other: Clinical assessment
Behavioral: questionnaires
Other: pulmonary function test
Biological: blood test
Biological: microbiology
Biological: histology
Other: imaging

SUMMARY:
Chronic inflammatory pulmonary diseases including chronic obstructive pulmonary disease (COPD), interstitial lung diseases (ILD), bronchiectasis, and cystic fibrosis (CF) are characterized by lung inflammation and remodelling. Clinical, functional, microbiological, biological, pathological and prognosis features are highly variable and heterogeneous. A precise phenotyping is a key-element to better understanding the pathophysiology of these chronic inflammatory diseases and to develop innovative treatment strategies.

The objectives of this prospective study is to analyze the clinical, demographic, biological, morphological, pathological, and microbiological characteristics in a cohort of patients diagnosed with COPD, ILD, bronchiectasis, and CF. The associations between clinical, demographic, biological, morphological, pathological, and microbiological features will be assessed.

The Cohort for Research and Innovation in Chronic Inflammatory Respiratory Diseases (the RINNOPARI Project: Recherche et Innovation en Pathologie Respiratoire Inflammatoire) is a monocentric study conducted at the University Hospital of Reims, France. Adult patients (>18 year-old) followed at the University Hospital of Reims and diagnosed with COPD, ILD, bronchiectasis, or CF will be considered for inclusion. Patients will sign an informed consent for inclusion. Exclusion criteria include "subjects protected by the law" as required by the French authorities. Control patients with no respiratory diseases after clinical and pulmonary function tests assessment will be also included. The expected number of patients included is 225 (COPD, n=100; CF, n=25; bronchiectasis, n=25; ILD, n=25; controls, n=50). Inclusion will be conducted for 36 months from September 2016 (9/30/2016) to September 2019 (9/30/2019).

For all COPD, ILD, bronchiectasis, and CF patients included, data will be registered at inclusion, and at follow-up visits for 10 years. Patients will be followed-up as usual care with no specific therapeutic intervention. For control patients, data will be registered at inclusion with no follow-up.

Data will be registered in a centralized anonymized database. The characteristics of the patients will be described as mean and standard deviation for quantitative data and as number and percentages for qualitative data. Comparisons and associations between groups and variables will be analyzed by Student, Wilcoxon, Chi2, Fischer exact, and Spearman tests as applicable. A p<0.05 will be considered as significant.

This study should help to better characterize clinical, demographic, biological, morphological, pathological, and microbiological characteristics and phenotypes in chronic inflammatory respiratory diseases.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 year-old) with COPD, CF, bronchiectasis or ILD

Exclusion Criteria:

* <18 year-old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2016-11-15 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2036-11 (Estimated)

PRIMARY OUTCOMES:
Specific measurements: cytokines (Th1, Th2, Th17, Tc1, Tc2, Tc17) measurements in blood sample | baseline
Specific measurements: cytokines (Th1, Th2, Th17, Tc1, Tc2, Tc17) measurements in blood sample | up to 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Derived] Charon L, Launois C, Perotin JM, Ravoninjatovo B, Mulette P, Ancel J, Guillard T, Muggeo A, Dormoy V, Griffon M, Carre S, Lebargy F, Deslee G, Dury S. Current cough and sputum assessed by the cough and sputum assessment-questionnaire (CASA-Q) is associated with quality of life impairment in cystic fibrosis. BMC Pulm Med. 2023 Nov 21;23(1):457. doi: 10.1186/s12890-023-02701-3. PMID 37990322
- [Derived] Dury S, Perotin JM, Ravoninjatovo B, Llerena C, Ancel J, Mulette P, Griffon M, Carre S, Perrin A, Lebargy F, Deslee G, Launois C. Identifying specific needs in adult cystic fibrosis patients: a pilot study using a custom questionnaire. BMC Pulm Med. 2021 Aug 18;21(1):270. doi: 10.1186/s12890-021-01613-4. PMID 34404378
- [Derived] Mulette P, Ravoninjatovo B, Guguen C, Barbe C, Ancel J, Dury S, Dumazet A, Perdu D, Perotin JM, Guillard T, Lebargy F, Deslee G, Launois C. Insomnia in adults with cystic fibrosis: strong association with anxiety/depression and impaired quality of life. BMC Pulm Med. 2021 Apr 1;21(1):108. doi: 10.1186/s12890-021-01473-y. PMID 33794842